CLINICAL TRIAL: NCT04698317
Title: Biodegradable Gelatin Sponge Loaded With Beta-Tricalcium Phosphate Sponges Incorporating Concentrated Growth Factors in the Treatment of Intra-bony Pocket Randomized Clinical and Radiographic Study
Brief Title: Beta-Tricalcium Phosphate and Concentrated Growth Factors in Treatment of Intra-bony Defect Randomized Clinical Trial
Acronym: RCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, malak mohamed shoukheba, associate prof., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ≤ ≥ ° ± µ ™ ®
Record Dates: First submitted 2020-12-31; First posted 2021-01-06 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Chronic Periodontitis; Intrabony Periodontal Defect; Concentrated Growth Factors
Keywords: Beta-Tricalcium Phosphate; regeneration; concentrated growth factors
MeSH Terms: conditions — Chronic Periodontitis | interventions — beta-tricalcium phosphate

STUDY DESIGN:
Intervention Model Description: 40 Patients will be randomly assigned to either test or control group. 20 patients will be treated by surgery plus biodegradable gelatin/beta-tricalcium phosphate sponges alone.
  (control group), the other 20 patients will be treated with the same surgical technique plus biodegradable gelatin sponge loaded with Beta-tricalcium phosphate socked in concentrated growth factors (test group).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- beta-tricalcium phosphate plus concentrated growth factors (Experimental): surgery plus biodegradable gelatin sponge loaded with Beta-tricalcium phosphate socked in concentrated growth factors (test group).
  Interventions: Procedure: open flap debridement; Other: use of Biodegradable Gelatin Sponge loaded with Beta-tricalcium Phosphate plus concentrated growth factors
- beta tricalcium phosphate alone(control group) (Placebo Comparator): surgery plus biodegradable gelatin/beta-tricalcium phosphate sponges alone. (control group),
  Interventions: Procedure: open flap debridement; Other: use of Biodegradable Gelatin Sponge loaded with Beta-tricalcium Phosphate alone

INTERVENTIONS:
Procedure: open flap debridement — Open flap for removal of diseased periodontal tissues and necrotic cementum
  Other Names: periodontal surgery
Other: use of Biodegradable Gelatin Sponge loaded with Beta-tricalcium Phosphate plus concentrated growth factors — use of Biodegradable Gelatin Sponge loaded with Beta-tricalcium Phosphate incorporating Concentrated Growth Factors in Periodontal Defect
  Other Names: regenerative surgery
  Arms: beta-tricalcium phosphate plus concentrated growth factors
Other: use of Biodegradable Gelatin Sponge loaded with Beta-tricalcium Phosphate alone — use of Biodegradable Gelatin Sponge loaded with Beta-tricalcium Phosphate alone in the Intrabony Periodontal Defect
  Other Names: Regenerative surgery
  Arms: beta tricalcium phosphate alone(control group)

SUMMARY:
This clinical study aimed to evaluate the efficacy of biodegradable gelatin sponge loaded with Beta-tricalcium phosphate socked in concentrated growth factors in the treatment of periodontal intra-bony defects, as compared with biodegradable gelatin/beta-tricalcium phosphate sponges alone.

DETAILED DESCRIPTION:
40 intra-bony defects in 40 patients will be selected from outpatient clinic of Oral Periodontology Clinic Faculty of Dentistry, Tanta University to participate in this study. Each defect had intra-bony depth > or = 4 mm and probing pocket depth (PPD) > or = 6 mm. Patients will be randomly assigned to either test or control group. 20 patients will be treated by surgery plus biodegradable gelatin/beta-tricalcium phosphate sponges alone.

(control group), the other 20 patients will be treated with the same surgical technique plus biodegradable gelatin sponge loaded with Beta-tricalcium phosphate socked in concentrated growth factors (test group).

Gingival index (GI), bleeding on probing, Probing pocket depth and clinical attachment level (CAL) will assessed at baseline, 3, and 6 months at the site to be treated. Cone beam radiographs evaluation will be taken at baseline, and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy patients were selected
* patients who had not received any medications for the previous six months that may interfere with periodontal tissue health or healing.
* Patients should demonstrate their ability to maintain good oral hygiene

Exclusion Criteria:

* Smokers and pregnant patients.
* Medically compromised patients and systemic conditions precluding periodontal surgery.
* Subjects who do not comply with oral hygiene measures as evidenced in recall visits.
* Sites with tooth mobility
* Restoration or caries in the site to be treated or non-vital tooth
* Restoration or caries in the site to be treated or non-vital tooth

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
gingival index | 6months
  gingival index will be recorded at baseline, 3, and 6 months at the site to be treated
bleeding on probing | 6 months
  bleeding on probing will be recorded at baseline, 3, and 6 months at the site to be treated
probing pocket depth | 6 months
  probing pocket depth will be recorded at baseline, 3, and 6 months at the site to be treated
clinical attachment level | 6 months
  clinical attachment level will be recorded at baseline, 3, and 6 months at the site to be treated
cone beam x ray measuring defect area | 6 months
  defect area will be recorded at baseline, and 6 months at the site to be treated
cone beam x ray measuring bone density | 6 months
  bone density will be recorded at baseline, and 6 months at the site to be treated

CONTACTS AND LOCATIONS:
Overall Officials: malak m shoukheba, Principal Investigator — Cairo University
Locations (1):
- Malak Mohamed Shoukheba, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No